CLINICAL TRIAL: NCT06626932
Title: Implications of Biological and Procedural Factors of 18-f FDG PET/CT Uptake by Normal Organs and Neoplastic Lesions
Brief Title: Implications of Biological and Procedural Factors of 18-f FDG Uptake by Normal Organs and Neoplastic Lesions
Status: Not yet recruiting | Type: Observational
Sponsor: mahenoor alaa eldeen naem (Other)
Responsible Party: Sponsor-Investigator, mahenoor alaa eldeen naem, Doctor, Assiut University
Organization: Assiut University (Other)
Other Study IDs: 18-FDG PET/CT scan
Record Dates: First submitted 2024-09-27; First posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-09

CONDITIONS: Oncologic Diseases
Keywords: 18-f FDG PET/CT
MeSH Terms: interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Radiation: 18 FDG (Fludeoxyglucose 18F) — 18-f FDG

SUMMARY:
To evaluate implications of biological and procedural factors of 18-f FDG PET/CT uptake on normal organs and neoplastic lesions.

DETAILED DESCRIPTION:
18-f FDG is used on oncological patients undergoing PET/CT study at our nuclear medicine unit , its uptake by the tissues depends on glucose blood level and consumption then we evaluate the implications of biological and procedural factors on the uptake by normal organs and neoplastic lesions using standardized uptake values SUVmax , mean and peak.

ELIGIBILITY:
Inclusion Criteria:

* cancer patients referred to nuclear medicine unit

Exclusion Criteria:

* patients with increased FDG uptake associated with non malignant causes such as diffuse bone marrow FDG uptake or lung infection or patients with extensive metastasis in target organs

Ages: 1 Year to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all cancer patients
Sampling Method: Probability Sample
Enrollment: 259 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
PET/CT scan on cancer patient will be performed to evaluate the biological and procedural factors of 18-f FDG uptake by multiple normal organs and neoplastic lesions using Standardized uptake values | 2 years
  SUV mean , suv peak and suv max

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Asyut, Egypt